CLINICAL TRIAL: NCT04225598
Title: Emergency Department-Initiated Buprenorphine Validation Network Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); The Emmes Company, LLC (Industry); Harvard Medical School (HMS and HSDM) (Other); University of Pennsylvania (Other); NYU Langone Health (Other); Icahn School of Medicine at Mount Sinai (Other); Alameda Health System (Other); Weill Medical College of Cornell University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000026164; 2UG1DA015831-19 (NIH)
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Opioid-use Disorder
Keywords: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XR-BUP (Experimental): Injectable buprenorphine
  Interventions: Drug: CAM2038
- Standard SL-BUP (Active Comparator): Sublingual buprenorphine
  Interventions: Drug: Buprenorphine Sublingual Product

INTERVENTIONS:
Drug: CAM2038 — Patients will receive a 24 mg dose of injectable CAM2038 in the ED on Day 0.
  Arms: XR-BUP
Drug: Buprenorphine Sublingual Product — COWS ≥ 8: Patients will receive 4mg of SL-BUP for a COWS score of 8-12 (mild withdrawal). After 30-45 minutes if tolerated and no unanticipated adverse reactions, an additional 4mg can be administered for a total of 8mg in the ED. Patients presenting with moderate-severe withdrawal (COWS >≥ 13) will receive an initial dose of 8mg SL-BUP. All patients will receive a buprenorphine prescription and instructions for additional BUP doses to allow for up to a dose of 12mg if needed, and for 16mg each subsequent day until their scheduled follow up appointment for ongoing MOUD (medications for opioid use disorder).
  COWS 4-7: Patients will be provided with a uniform set of instructions to guide unobserved (home) induction. They will be prescribed doses of SL-BUP to allow them to take dose up to 12mg in the 24 hours after discharge. All patients will also receive a buprenorphine prescription for 16mg each subsequent day until their scheduled follow up appointment for ongoing MOUD.
  Arms: Standard SL-BUP

SUMMARY:
This study will (1) recruit, train and provide resources to approximately 30 Emergency Department (ED) sites throughout the U.S. using implementation facilitation strategies to provide ED-initiated buprenorphine (BUP) for patients presenting with opioid use disorder (OUD) who are not receiving medications for opioid use disorder (MOUD). Once implementation is adequately achieved, the sites will (2) conduct a randomized controlled trial (RCT) to compare the effectiveness of sublingual buprenorphine (SL-BUP) versus extended-release buprenorphine (XR-BUP) on ED patients' engagement in formal addiction treatment 7-days after their ED visit. In addition, in an ancillary component of the study, the investigators will (3) assess the use of XR-BUP in ED patients with Clinical Opioid Withdrawal Scale (COWS) scores < 8 in a case series to potentially expand the eligibility of patients in the larger RCT to those presenting with little to no opioid withdrawal symptoms. Finally, the investigators will (4) develop and validate ED electronic health record (EHR) opioid-related phenotypes, both of which will inform the main RCT.

DETAILED DESCRIPTION:
The study will be comprised of four components as outlined below:

1. Site implementation component:

   In this component, the investigators will use previously developed implementation facilitation strategies and resources to train ED providers and staff at approximately 30 diverse EDs in treatment initiation with SL-BUP and XR-BUP and develop ED buprenorphine protocols and procedures. The investigators anticipate that this will result in a minimum of 24 sites (80%) that will meet the implementation milestones for competence in ED-initiated BUP using standard SL and XR-BUP inductions.
2. Effectiveness RCT component:

   This component is a large pragmatic RCT using a Hybrid Type 1 Effectiveness-Implementation design. Sites that satisfactorily complete the site implementation component will be activated on a rolling basis for the RCT after demonstrated implementation milestones have been met. In this Hybrid Type 1 design the primary research question is the effectiveness of SL-BUP induction compared with that of XR-BUP on the primary outcome measure of engagement in formal addiction treatment at 7-days post ED visit. This design also allows us to gather information and report on implementation processes.
3. Ancillary component - XR-BUP Induction for patients with COWS < 8:

   This observational case series will begin in advance of the Effectiveness RCT component at approximately 4 ED sites with extensive experience in ED-initiated BUP. The investigators will collect quantitative and qualitative data on the use of XR-BUP in ED patients with low COWS scores for approximately 75 patients. Sites will receive a supply of XR-BUP for provision to up to 5 patients with a COWS score > 8. The purpose is to pre-study the procedures at the four ancillary study sites on treating OUD patients with XR-BUP prior to initiation of the ancillary component. Data collected from this pre-study will not be included in the analysis of the ancillary and effectiveness RCT component. These initial up to 20 pre-study patients will meet all other study criteria and undergo all assessments. It is anticipated that the information collected from the 75 patients in the ancillary component will allow for modification to the larger Effectiveness RCT by expanding eligibility criteria to include patients with COWS <8.
4. Development and validation of EHR ED opioid-related phenotypes component:

   In this component, the investigators will develop EHR phenotypes of opioid-related illnesses that accurately and automatically characterize patient conditions, enhance the ability to actively monitor and surveil, and better identify representative samples and patients potentially eligible for study inclusion, leading ultimately to an enhanced inclusion and understanding of opioid-related conditions. At the primary Yale New Haven Health System sites, the phenotypes (rules- and machine learning-based) will be iteratively developed and internally validated. The rules-based phenotype will be mapped to a common data model and externally validated at 4 trial sites.
5. An exploratory outcome of this study will be to assess the impact of COVID-19 on ED use for opioid-related diagnoses using EHR data.

The primary focus of this clinicaltrials.gov registration are the RCT outcomes. Implementation and ancillary outcomes will be identified as secondary outcomes for the purpose of this clinicaltrials.gov registration

ELIGIBILITY:
RCT Component:

Inclusion Criteria:

1. Be 18 years or older
2. Treated in the ED during study screening hours
3. Meet DSM-5 (Diagnostic and Statistical Manual) diagnostic criteria for moderate to severe OUD
4. Have a COWS score of > or equal to 4
5. Have a urine toxicology test that is positive for opioids (opiates, oxycodone, buprenorphine). Patients with urines that are only positive for fentanyl will be eligible if their clinical history and physical exam are consistent with opioid use and they meet DSM-5 criteria for moderate to severe OUD.
6. Able to speak English sufficiently to understand the study the study procedures and provide written informed consent to participate in the study. (Exception may be made if sites with large population of Spanish speaking patients are accepted for participation in the study and study materials are translated into Spanish. Translated study materials will be reviewed and approved by the Institutional Review Board) IRB of record prior to use.)

Exclusion Criteria:

1. Have urine toxicology test that is positive for methadone
2. Be pregnant as determined by human chorionic gonadotropin (hCG) testing at the index ED visit
3. Have a medical or psychiatric condition that requires hospitalization
4. Opioid administration (excluding BUP) at the index ED visit, prior to enrollment, and COWS remains < 8 during ED stay
5. Be actively suicidal or severely cognitively impaired precluding informed consent
6. Present from an extended care facility (e.g., skilled nursing facility)
7. Require continued prescription opioids for a pain condition
8. Be a prisoner or in police custody at the time of index ED visit
9. Be currently (anytime within the past 14 days) enrolled in formal addiction treatment, including by court order. Patients enrolled in formal addiction who are not receiving MOUD are eligible
10. Be unable to provide reliable locator information including 2 contact numbers in addition to their own
11. Be unwilling to follow study procedures (e.g., unwilling to provide permission to contact referral provider/program or unavailable for the follow-up assessments)
12. Have prior enrollment in the current study component

Ancillary Component:

Inclusion Criteria:

1. Be 18 years or older
2. Treated in the ED during study screening hours
3. Meet DSM-5 diagnostic criteria for moderate to severe opioid use disorder
4. Have a COWS <8
5. Have a urine toxicology test that is positive for opioids (opiates, oxycodone, or buprenorphine). Patients with urines that are only positive for fentanyl on the point of care test strip will be eligible if their clinical history and physical exam are consistent with opioid use and they meet DSM-5 criteria for moderate to severe OUD.
6. Be able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

1. Have a urine toxicology test that is positive for methadone
2. Be pregnant as determined by human chorionic gonadotropin (hCG) testing at the index ED visit
3. Have a medical or psychiatric condition that requires hospitalization at the index ED visit, prior to enrollment
4. Be actively suicidal or severely cognitively impaired precluding informed consent
5. Present from an extended care facility (e.g., skilled nursing facility)
6. Require continued prescription opioids for a pain condition
7. Be a prisoner or in police custody at the time of index ED visit
8. Be currently (anytime within the past 7 days) enrolled in formal addiction treatment, including by court order. Patients enrolled in formal addiction treatment but are not receiving MOUD are eligible
9. Be unable to provide reliable locator information including 2 contact numbers in addition to their own
10. Be unwilling to follow study procedures (e.g., unwilling to provide permission to answer daily assessments until day 7)
11. Have prior enrollment in the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
RCT Component: Patient engagement (yes/no) in formal addiction treatment at 7 days post randomization | 7 days post randomization
  Engagement in formal addiction treatment will be defined as enrollment and receiving formal addiction treatment on the 7th day post randomization, confirmed by contact with the facility and/or treating clinician. Formal addiction treatment will be operationally defined as those treatments consistent with the American Society of Addiction Medicine's levels of care (1-4) and can include a range of clinical settings including office-based providers of BUP or naltrexone, opioid treatment programs (OTPs), intensive outpatient, inpatient, or residential treatments. Patients do not need to be receiving MOUD at 7 days to be considered engaged in formal addiction treatment. Participation in a mutual-help program such as Alcoholics Anonymous (AA) or (Narcotics Anonymous) NA alone will not be considered as engagement in formal addiction treatment. Additional analyses evaluating the effects of patient and site characteristics will also be conducted.

SECONDARY OUTCOMES:
RCT Component: Engagement in MOUD (yes/no) at 7 days post randomization | 7 days post randomization
  self-report verified with treatment provider(s)
RCT Component: Patient engagement (yes/no) in formal addiction treatment at 30 days post randomization | 30 days post randomization
  Engagement in formal addiction treatment will be defined as enrollment in formal addiction treatment on the 30th day post randomization, confirmed by direct contact with the facility and/or treating clinician. Formal addiction treatment will be operationally defined as those treatments consistent with the American Society of Addiction Medicine's levels of care (1-4) and can include a range of clinical settings including office-based providers of BUP or naltrexone, OTPs, intensive outpatient, inpatient, or residential treatments. Patients do not need to be receiving MOUD on the 30th day post randomization to be considered engaged in formal addiction treatment. Participation in a mutual-help program such as Alcoholics or Narcotics Anonymous alone will not be considered as engagement in formal addiction treatment. Additional analyses evaluating the effects of patient and site characteristics will also be conducted.
RCT Component: Patient Engagement in MOUD (yes/no) at 30 days post randomization | 30 days post randomization
  self report verified with treatment provider(s)
RCT Component: Self-reported days of illicit opioid use (past 7 days) at 7 days post randomization | 7 days post randomization
  The Timeline Follow-back procedure will be used to elicit the patient participant's self-reported days of use of opioids.
RCT Component: Self-reported days of illicit opioid use (past 7 days) at 30 days post randomization | 30 days post randomization
  The Timeline Follow-back procedure will be used to elicit the patient participant's self-reported days of use of opioids.
RCT Component: Craving scores at 7 days post randomization | 7 days post randomization
  The investigators will use visual analogue scales (VAS) to assess craving, desire to use opioids and need to use opioids with a scale of 0-100.
RCT Component: Healthcare services utilization (past 30 days) regarding ED visits and hospitalizations at 30 days post randomization | 30 days post randomization
  A brief, structured interview regarding health care utilization (inpatient and outpatient) will be used, which collects information on the type and amount of services received. This includes ED visits, hospitalizations, primary medical care visits (excluding those for BUP treatment and self-help sources of support (e.g., NA).
RCT Component: Patient satisfaction with BUP at 7 days post randomization | 7 days post randomization
  The investigators will modify the patient satisfaction scale where overall experience is rated from 1 to 5 (1 is completely ineffective and 5 is completely effective) and treatment characteristics are rated 1 to 7 (1 is not important and 7 is extremely important) based on previous published data.
RCT Component: Overdose Events at 30 days post randomization | 30 days post randomization
  Assessment of past 30-day overdose events will be completed at 30 days post study enrollment. In addition, Site PIs will search local electronic medical records for fatal and non-fatal overdose events.
Ancillary Component: Proportion of participants that experience a 5 or greater increase in COWS score within 4 hours of of XR-BUP administration | Within 4 hours of XR-BUP administration
  Clinical Opiate Withdrawal Scale (COWS) - the COWS is a validated measure of the severity of opioid withdrawal that consists of 11 subjective and objective items. Scores on the individual items are combined to a single overall score that has been used to determine the SL-BUP induction strategy. COWS scoring, and interpretation is as follows: Score: 5-12 = mild opioid withdrawal; 13-24 = moderate opioid withdrawal; 25-36 = moderately severe opioid withdrawal; more than 36 = severe opioid withdrawal.
Ancillary Component: Proportion of participants that transition to moderate withdrawal (COWS 13-24) within 4 hours of XR-BUP administration | Within 4 hours of XR-BUP administration
  Clinical Opiate Withdrawal Scale (COWS) - the COWS is a validated measure of the severity of opioid withdrawal that consists of 11 subjective and objective items. Scores on the individual items are combined to a single overall score that has been used to determine the SL-BUP induction strategy. COWS scoring, and interpretation is as follows: Score: 5-12 = mild opioid withdrawal; 13-24 = moderate opioid withdrawal; 25-36 = moderately severe opioid withdrawal; more than 36 = severe opioid withdrawal.
Ancillary Component: Proportion of participants that experience clinician determined precipitated withdrawal within 1 hour of XR-BUP administration | Within 1 hour post XR-BUP injection
  Assessment of Proportion of participants that experience clinician determined precipitated withdrawal within 1 hour of XR-BUP administration.

OTHER OUTCOMES:
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): Engagement | 7 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): QALYs | 7 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): Abstinent Years | 7 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): Engagement | 30 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): QALYs | 30 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.
RCT Component: Cost effectiveness of XR-BUP compared to SL-BUP using ICER (incremental cost-effectiveness ratio): Abstinent Years | 30 days post randomization
  The final outcome measure for the cost-effectiveness analysis is the ICER (incremental cost-effectiveness ratio), which includes the relevant cost differential between the study arms in the numerator, and the difference in a chosen effectiveness measure in the denominator. 3 types of ICERs will be generated, each one with a different effectiveness measure (engagement in formal addiction treatment at 30 days; quality-adjusted life-years (QALYs) gained; and Abstinent Years). The reason being that different ICERs are more relevant to certain potential stakeholder groups than others.

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Yale School of Medicine, Department of Emergency Medicine; David Fiellin, MD, Principal Investigator — Yale School of Medicine, Department of Internal Medicine
Locations (35):
- United States (35):
  - Highland Hospital, Oakland, California
  - San Leandro Hospital, San Leandro, California
  - Yale New Haven Health (Yale New Haven Hospital), New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Presybterian Hospital, Albuquerque, NM, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Bellevue Hospital, New York, New York
  - Icahn School of Medicine, New York, New York
  - Columbia University Irving Medical Center- NY Presbyterian, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Pennsylvania Presbyterian Medical Center/Hospital of UPENN, Philadelphia, Pennsylvania
  - Temple University Hospital - Episcopal Campus, Philadelphia, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital/The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Washington Medical Center- Harborview/Montlake, Seattle, Washington
  - West Virginia University - Berkeley Medical Center, Martinsburg, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
In line with the National Institutes of Health Helping to End Addiction Long-term (NIH HEAL) Initiative Public Access and Data Sharing Policy, publications and underlying primary data will be made available to the public.
Time Frame: Data will be made available after 1) the primary paper has been accepted for publication, or 2) the data is locked for more than 18 months, whichever comes first.

REFERENCES:
- [Derived] D'Onofrio G, Herring AA, Hawk KF, Perrone J, Cowan E, McCormack RP, Dziura J, Matthews AG, Pantalon MV, Owens P, Martel S, Coupet E Jr, Lofwall MR, Walsh SL, Edelman EJ, Carpenter JE, Strout TD, Baumann MR, Anderson E, Barrett TW, Dorey A, Taillac P, Cochran G, Crandall CS, Wilson J, Manteuffel J, Cole JB, Whiteside LK, Jones C, Samuels E, Huntley K, Fiellin DA; ED INNOVATION Investigators. Emergency Department-Initiated Buprenorphine for Opioid Use Disorder: A Randomized Clinical Trial. JAMA. 2026 Feb 11. doi: 10.1001/jama.2025.27019. Online ahead of print. PMID 41670966
- [Derived] D'Onofrio G, Herring AA, Perrone J, Hawk K, Samuels EA, Cowan E, Anderson E, McCormack R, Huntley K, Owens P, Martel S, Schactman M, Lofwall MR, Walsh SL, Dziura J, Fiellin DA. Extended-Release 7-Day Injectable Buprenorphine for Patients With Minimal to Mild Opioid Withdrawal. JAMA Netw Open. 2024 Jul 1;7(7):e2420702. doi: 10.1001/jamanetworkopen.2024.20702. PMID 38976265
- [Derived] Snavely AC, Paradee BE, Ashburn NP, Allen BR, Christenson R, O'Neill JC, Nowak R, Wilkerson RG, Mumma BE, Madsen T, Stopyra JP, Mahler SA. Derivation and validation of a high sensitivity troponin-T HEART pathway. Am Heart J. 2023 Feb;256:148-157. doi: 10.1016/j.ahj.2022.11.012. Epub 2022 Nov 16. PMID 36400184